CLINICAL TRIAL: NCT01907178
Title: Assessment of Postoperative Pain Management in Patients Undergoing Total Knee Arthroplasty Immediately After Surgery and Following Discharge From Hospital.
Brief Title: Postoperative Pain Management in Hospital and Following Discharge From Hospital.
Status: Completed | Type: Observational
Sponsor: Trinity Health Of New England (Other)
Responsible Party: Sponsor
Other Study IDs: 13-06-002
Record Dates: First submitted 2013-06-28; First posted 2013-07-24 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Arthropathy of Knee Joint
Keywords: total knee arthroplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Postoperative pain management: The postoperative pain level will be assessed during hospitalization and at home, in patients undergoing total knee replacement

SUMMARY:
To investigate postoperative pain management in patients undergoing knee or hip replacement while they are in the hospital and following discharge to their home. Additionally, sample questions will be asked prior to surgery to predict patient's postoperative pain experience.

DETAILED DESCRIPTION:
We hypothesize that patients experience more postoperative pain at home than they do in hospital and factors such as preoperative anxiety, depression, and preoperative pain affect the level of postoperative pain experienced by patients. A total of 200 patients undergoing total knee surgery will be enrolled in this observational study. They will be asked to fill a baseline questionnaire including demographic information, medical problems, anxiety, depression, preoperative pain level, etc. Following routine standard anesthesia and surgery, patient's pain will be assessed every 4 hours when they are in the hospital after surgery, then daily assessment for 1 week after they are discharged home followed at 2 months, and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total knee arthroplasty

Exclusion Criteria:

* Patients attending rehabilitation facilities after discharge
* unwilling or unable to provide consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated at Saint Francis Hospital undergoing total knee replacement
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06-16 (Actual); Study Completion 2015-06-16 (Actual)

PRIMARY OUTCOMES:
Pain scores | during hospital stay (average 3 days)
  Pain scores (at rest & with exercise) will be collected during the hospital stay

SECONDARY OUTCOMES:
preoperative anxiety scores | preoperative
  Analysis of preoperative anxiety scores.
Preoperative depression scores | preoperative
  Analysis of preoperative depression score.

OTHER OUTCOMES:
Pain medication consumption | during hospital stay (average 3 days)
  pain medication consumption will be collected during hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Sinha, MD, Principal Investigator — Saint Francis Hospital
Locations (1):
- Saint Francis Hospital and Medical Center, Hartford, Connecticut, United States